CLINICAL TRIAL: NCT04197570
Title: Opioid-free Anesthesia for Open Cardiac Surgery: A Prospective Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB19-024
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Opioid Use; Heart; Surgery, Heart, Functional Disturbance as Result; Anesthesia
Keywords: Opioid Free Anesthesia; Cardiac Surgery; Non-opioid Anesthesia; Dexmedetomidine; Hemodynamic; Opioid; Fentanyl; Cardiac Anesthesia; Cardiopulmonary Bypass; post sternotomy pain
MeSH Terms: interventions — Analgesics, Non-Narcotic

STUDY DESIGN:
Intervention Model Description: The investigators plan to enroll 158 subjects at Virginia Mason Medical Center that are undergoing open cardiac surgery. Subjects who volunteer to be involved in the study will be randomized to either the opioid free or traditional anesthetic arm. Subjects will be blinded to the assigned arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-based anesthetic (Active Comparator): Premedication
  -midazolam 2mg IV x 1 as need for anxiety, at the discretion of the anesthesiologist
  Induction
  * Fentanyl 2-4 mcg/kg IV bolus
  * Propofol 1-3 mg/kg IV
  * Paralytic and vasoactive medications at the discretion of the anesthesiologist
  Maintenance
  * Fentanyl 1-2 mcg/kg IV bolus immediately prior to sternotomy & aortic cannulation
  * Fentanyl 1-2mcg/kg IV bolus immediately following removal of bypass cannula
  * Dexmedetomidine 0.4 mcg/kg/hr IV infusion
  * Isoflurane titrated at the discretion of the anesthesiologist
  * Vasoactive medications at the discretion of the anesthesiologist for hemodynamic management
  During chest closure:
  * start Propofol 25-75mcg/kg/min IV infusion
  * continue dexmedetomidine 0.4mcg/kg/hr IV infusion
  * titrate off isoflurane
  * Acetaminophen 1000mg IV
  Interventions: Drug: Opioid Anesthetics
- Opioid-free anesthetic (Experimental): Premedication
  -midazolam 2mg IVx1 as needed for anxiety, at the discretion of the anesthesiologist
  Induction
  * Dexmedetomidine 1mcg/kg IV
  * Propofol 1-3mg/kg IV
  * Paralytic and vasoactive medications at the discretion of the anesthesiologist
  Maintenance
  * Dexmedetomidine 0.8-1.0 mcg/kg/hr IV infusion
  * Isoflurane titrated at the discretion of the anesthesiologist
  * May add propofol infusion if clinically indicated
  * Vasoactive medications at the discretion of the anesthesiologist for hemodynamic management
  During chest closure:
  * start Propofol 25-75mcg/kg/min IV infusion
  * continue dexmedetomidine 0.4 - 1.0 mcg/kg/hr IV infusion
  * titrate off isoflurane
  * Acetaminophen 1000mg IV
  Interventions: Drug: Non Opioid Analgesics

INTERVENTIONS:
Drug: Opioid Anesthetics — see arm/group description
  Other Names: Opioid-based anesthetic
  Arms: Opioid-based anesthetic
Drug: Non Opioid Analgesics — see arm/group description
  Other Names: Opioid-free anesthetic
  Arms: Opioid-free anesthetic

SUMMARY:
This study will compare an opioid free anesthetic, using dexmedetomidine, to a traditional opioid based anesthetic, using fentanyl, for patients undergoing cardiac surgery with regards to hemodynamic stability in the first 10 minutes after induction.

DETAILED DESCRIPTION:
This is a single center, blinded, prospective, randomized controlled trial. A total of 158 subjects (79 subjects in each arm) are planned. The control group will receive a traditional cardiac anesthetic using opioids, for which induction will include fentanyl and propofol. The experimental arm will receive an opioid free anesthetic with an induction bolus of dexmedetomidine and propofol. The investigators hypothesize that using the opioid free technique will be more hemodynamically stable within the first 10 minutes of induction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at the time of consent.
* Undergoing non-emergent open cardiac procedures requiring cardiopulmonary bypass support, including: CABG, aortic aneurysm repair, valve repair/replacement, or CABG in combination with valve repair/replacement.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Chronic opioid use defined as preoperative MED >100 daily.
* Hypersensitivity or contraindication to any of the study medications.
* Pre-existing Alzheimer's/vascular dementia.
* Pre-existing psychiatric disorder precluding ability to provide informed consent or use a visual analogue scale for pain.
* Childs-Pugh Class C liver failure or acute liver failure.
* Emergent open heart surgery, including type A aortic dissections, trauma, or conversion (bail out) from another procedure such as cardiac catheterization, ablation, transcatheter aortic valve replacement or any other general surgical procedure.
* Pregnancy or lactating.
* Inability to comply with the requirements of the study, per investigator judgment.
* Patients determined to need an awake intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Mean arterial blood pressure-time integral | 10 minutes
  The primary endpoint is the area under the baseline mean arterial pressure (MAP) over the first 10 minutes after induction, called the MAP-time integral.

SECONDARY OUTCOMES:
Blood pressure variability pre-cardiopulmonary bypass | 2 hours
  highest and lowest blood pressure from induction to start of bypass
Heart rate variability pre-cardiopulmonary bypass | 2 hours
  highest and lowest heart rate from induction to start of bypass
Vasopressor usage intra- and post-operatively | 18 hours
  Number of vasopressors and doses from induction to start of cardiopulmonary bypass, leaving operating room and 12 hours postop
Arrhythmias or EKG changes | 14 days
  Intraoperative EKG changes or evidence of echocardiographic ischemia prior to heparin. Antiarrhythmic medications given intraoperative or in first 24 hours postop. New permanent pacemaker placed during hospital admission.
Delirium medications | 24 hours
  Delirium medications administered 24 hours after ICU admission
Delirium | 24 hours
  CAM-ICU scores at 12 hours and 24 hours after ICU admission
Postoperative pain scores | 24 hours
  Numerical Rating Scale Pain Scores (Range: 0-10, where 0 is no pain and 10 is the worst pain)
Opioid consumption | 24 hours
  Total opioid utilization 24hours postoperatively (morphine equivalent dose)
Postoperative nausea/vomiting | 24 hours
  Number of antiemetic doses administered
Time to extubation | 1-36 hours
  Time from arrival in ICU to extubation
ICU length of stay | 1-5 days
  Time from arrival in ICU to time of transfer order out of ICU
Hospital length of stay | 3-14 days
  Time begins day of surgery to day of discharge. Time in days
Reintubation or readmission to ICU | 0-14 days
  After being extubated or being transferred out of ICU
major adverse cardiovascular event or mortality | 30 days
  Major adverse cardiovascular event (eg., myocardial ischemia, stroke) or death
Postoperative pain questionnaire | 6 months
  30 day, 3 month and 6 month pain questionnaire as well as post-sternotomy opioid use (as determined by reviewing Washington PMP data). Numerical Rating Scale Pain Scores (Range: 0-10, where 0 is no pain and 10 is the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bain, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No